CLINICAL TRIAL: NCT00846716
Title: Exploratory Study to Investigate the Suppressive Effect of Oral Anti-Diabetic Drug (TZD) on Progression of Diabetic Nephropathy on
Brief Title: Shiga Progression of Diabetes, Nephropathy and Retinopathy
Acronym: SHIP-DINER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiga University (Other)
Collaborators: Kanazawa Medical University (Other); Nagahama Red Cross Hospital (Other); Nagahama City Hospital (Other); Kohka Public Hospital (Unknown); Second Okamoto General Hospital (Unknown); Omihachiman COmmunity Medical Center (Unknown); Yasu Hospital (Unknown); Toyosato Hospital (Unknown); Ako City Hospital (Other); Horide Clinic (Unknown); Kawabata Clinic (Unknown); Seta Clinic (Unknown); Shiga Clinic (Unknown); Osaka University (Other); NTT West Osaka Hospital (Unknown); Hyogo prefectural Amagasaki Hospital (Unknown); Tomita Clinic (Unknown); Sawada Clinic (Unknown); Social Insurance Shiga Hospital (Unknown)
Responsible Party: Atsunori Kashiwagi, Shiga University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008.9.18 ver2-4
Record Dates: First submitted 2008-12-11; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Diabetic Retinopathy; pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Diabetic Retinopathy | interventions — Biguanides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone add on to SU or biguanide (Experimental)
  Interventions: Drug: Pioglitazone add on to SU or biguanide
- SU or Biguanide (Active Comparator)
  Interventions: Drug: SU or Biguanide

INTERVENTIONS:
Drug: Pioglitazone add on to SU or biguanide — As an initial dosing, 15mg/day of pioglitazone is administered to the patients for 2 years, who are taking SU or biguanide.
  Arms: Pioglitazone add on to SU or biguanide
Drug: SU or Biguanide — As an initial dose,a common dose of SU or biguanide is administered to the patients for 2 years.
  Arms: SU or Biguanide

SUMMARY:
The purpose of this study is to investigate whether the oral anti-diabetic drug, Thiazolidine (TZD) is effective in suppression of onset or progressin of diabetic nephropathy in Japanese type 2 diabetic patients.

DETAILED DESCRIPTION:
2. Outcome measures:

1. Primary endpoint Onset or progression of diabetic nephropathy
2. Secondary endpoints (1)Progression of diabetes mellitus (2)Change in HbA1c (3)Change in albumin-creatinine ratio (4)Change in GFR (5)CHange in cystatin C

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Less than 8.0% in HbA1c
* Less than 300 mg/g Cr of urinary albumine level
* Concomitant therapy with SU and/or Biguanide
* Untreated hypertension and hypertension treated with ARB or ACEI

Exclusion Criteria:

* History of heart failure and concomitant heart failure
* History of administration of TZD agent
* Severe hepatic dysfunction with more than 3 times higher than upper limit of normal range of GOT, GPT or rGPT
* Severe renal dysfunction with more than 2.5 of Cr
* History of AE with TZD agent
* Insulin treatment
* Concomitant urinary track infection

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Onset and progression of diabetic nephropathy | 2 years

SECONDARY OUTCOMES:
Progression of diabetes mellitus change from the baseline in HbA1c change from the baseline in albumine/creatinine ratio change from the baseline in cystatin C onset and progression of diabetic retinopathy safety assessment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Atsunori Kashiwagi, PhD., Study Chair — Tsukiwa-machi, Seta, Otsu, Shiga, Japan
Locations (1):
- Shiga University of Medical Science, Ōtsu, Shiga, Japan